CLINICAL TRIAL: NCT05859880
Title: A Community-based Video-conference-delivered Expressive Writing Intervention for Caregivers of Persons With Cancer
Brief Title: Expressive Writing for Caregivers of Persons With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00017135
Record Dates: First submitted 2023-03-16; First posted 2023-05-16 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Quality of Life; Distress, Emotional

STUDY DESIGN:
Intervention Model Description: Waitlist control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active intervention (Experimental): Participants will attend four group-based expressive writing sessions led by a trained facilitator. All sessions will be delivered via videoconference. Sessions will occur weekly over the course of 4 consecutive weeks and will not exceed 60 minutes in length. Each session will include a 15- to 20-minute writing stint whereby participants are asked to write about their deepest thoughts and feelings regarding their loved one's cancer and their role as caregiver. All participants will be given a Rocketbook for this purpose, a spiral notebook that has the look and feel of a standard paper notebook but uses a pen with erasable ink. The writing stint will be followed by a group discussion; participants will be invited to share what they wrote about (if so desired) and their reactions to the writing process. Each session will end with a debriefing and erasure of the writing content just created. This will ensure privacy of the material and may be perceived as cleansing.
  Interventions: Behavioral: Expressive writing intervention
- Waitlist control (Placebo Comparator): Procedures are exactly the same as for the experimental arm but delayed.
  Interventions: Behavioral: Expressive writing intervention

INTERVENTIONS:
Behavioral: Expressive writing intervention — 4 videoconference-delivered group-based expressive writing sessions

SUMMARY:
The goal of this clinical trial is to test the effects of an expressive writing intervention for caregivers of persons with cancer. The main questions the study aims to answer are:

1. Does participation in a group-based, videoconference-delivered expressive writing intervention improve mood and quality of life for caregivers of persons with cancer?
2. Is greater improvement associated with writing that is more emotionally expressive or personally revealing, or with group-based sessions characterized by certain linguistic features such as greater emotionality?
3. Is benefit greater for certain subgroups of caregivers, such as those who are younger or who identify as female in gender?

Participants will be asked to join four videoconference-delivered, group-based expressive writing sessions. This will be done in groups of 4-8 caregivers and led by a trained facilitator. During each session, participants will write about their deepest thoughts and feelings about their loved one's cancer and their experiences as a caregiver. They will then discuss as a group any reactions to the writing process.

Participants will be randomly assigned to either active intervention (receiving the intervention as soon as a group is formed) or waitlist control. Researchers will compare active and waitlist control participants on to pre- to post-intervention changes in mood and quality of life.

DETAILED DESCRIPTION:
A diagnosis of cancer reverberates throughout the family. Family caregivers take on a wide range of responsibilities, such as monitoring medical symptoms, communicating with the patient's medical team, managing insurance claims, providing transportation, and assisting with activities of daily living. Psychological distress is common. Caregivers often feel unprepared for their role, and socially isolated from others. Physical impacts have also been documented, from fatigue to sleep disturbance to immune dysfunction. To alleviate some of these difficult sequelae of cancer caregiving, we propose to test the utility of a brief, low-cost, non-pharmacologic, behavioral intervention for persons providing care for a loved one with cancer. Specifically, we will test the effects of an expressive writing (EW) intervention. The basic paradigm asks participants to write for 20 minutes on four separate occasions about a trauma or stressor. Initial work conducted with undergraduate samples showed benefit of EW. Since then, EW studies have been conducted across a variety of populations including persons coping with chronic illness. Benefits have ranged from better lung function among asthmatics to fewer physical symptoms among women with breast cancer. One meta-analysis of 146 studies across 10,994 participants reported positive effect sizes (mental or physical health benefits) for 102 of the studies (70%). Notable gaps in this literature include testing with cancer caregivers (with some exceptions) and use of novel delivery formats.

Specific aims are: (1) To examine the effects of a group-based, videoconference-delivered EW program on emotional, social, and physical well-being among informal caregivers of persons diagnosed with cancer; (2) To identify social and linguistic mechanisms by which participation in the group-based EW intervention may improve distress; and (3) To identify potential moderators of benefit including age, gender identity, relationship to the patient, and baseline social constraints.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Self-identify as informal caregiver for an adult (age 18+) diagnosed with stage II-IV breast, ovarian, prostate, colon, rectal, or lung cancer within the past 2 years
* English speaking and comprehending
* Access to a desktop computer, laptop, tablet or smartphone and Wireless Fidelity (WIFI) to complete surveys and participate in videoconference-based expressive writing sessions

Exclusion Criteria:

-Caregiver for pediatric cancer patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2025-04-06 (Actual); Study Completion 2025-04-06 (Actual)

PRIMARY OUTCOMES:
Psychological distress | change from baseline psychological distress at 6 weeks
  Profile of Mood States, 2nd edition (0-4, higher values indicate greater distress)
Quality of life, general | change from baseline quality of life at 6 weeks
  World Health Organization Quality of Life - Abbreviated version (0-100, higher values indicate greater quality of life)
Quality of life, caregiver-specific | change from baseline caregiver-specific quality of life at 6 weeks
  Caregiver Quality of Life Index-Cancer (0-140, higher values indicate greater quality of life)

SECONDARY OUTCOMES:
Depression | change from baseline depression at 6 weeks
  Center for Epidemiologic Studies Depression-10 (0-30, higher values indicate greater depression)
Perceived stress | change from baseline perceived stress at 6 weeks
  Perceived Stress Scale (0-40, higher values indicate greater stress)

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Support Community Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available to other researchers
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of publication of study results
Access Criteria: Access will be provided on a case by case basis, after review of the requestor's proposed use for the data. Requests will be reviewed by the principal investigator and at least one other investigator.

REFERENCES:
- [Background] Glajchen M. The emerging role and needs of family caregivers in cancer care. J Support Oncol. 2004 Mar-Apr;2(2):145-55. PMID 15328817
- [Background] Jayani R, Hurria A. Caregivers of older adults with cancer. Semin Oncol Nurs. 2012 Nov;28(4):221-5. doi: 10.1016/j.soncn.2012.09.004. PMID 23107179
- [Background] Areia NP, Fonseca G, Major S, Relvas AP. Psychological morbidity in family caregivers of people living with terminal cancer: Prevalence and predictors. Palliat Support Care. 2019 Jun;17(3):286-293. doi: 10.1017/S1478951518000044. Epub 2018 Feb 26. PMID 29478419
- [Background] Geng HM, Chuang DM, Yang F, Yang Y, Liu WM, Liu LH, Tian HM. Prevalence and determinants of depression in caregivers of cancer patients: A systematic review and meta-analysis. Medicine (Baltimore). 2018 Sep;97(39):e11863. doi: 10.1097/MD.0000000000011863. PMID 30278483
- [Background] Northouse LL, Katapodi MC, Schafenacker AM, Weiss D. The impact of caregiving on the psychological well-being of family caregivers and cancer patients. Semin Oncol Nurs. 2012 Nov;28(4):236-45. doi: 10.1016/j.soncn.2012.09.006. PMID 23107181
- [Background] Girgis A, Lambert S, Johnson C, Waller A, Currow D. Physical, psychosocial, relationship, and economic burden of caring for people with cancer: a review. J Oncol Pract. 2013 Jul;9(4):197-202. doi: 10.1200/JOP.2012.000690. Epub 2012 Dec 4. PMID 23942921
- [Background] Teixeira RJ, Applebaum AJ, Bhatia S, Brandao T. The impact of coping strategies of cancer caregivers on psychophysiological outcomes: an integrative review. Psychol Res Behav Manag. 2018 May 24;11:207-215. doi: 10.2147/PRBM.S164946. eCollection 2018. PMID 29872357
- [Background] Stanton AL, Danoff-Burg S, Sworowski LA, Collins CA, Branstetter AD, Rodriguez-Hanley A, Kirk SB, Austenfeld JL. Randomized, controlled trial of written emotional expression and benefit finding in breast cancer patients. J Clin Oncol. 2002 Oct 15;20(20):4160-8. doi: 10.1200/JCO.2002.08.521. PMID 12377959
- [Background] Frattaroli J. Experimental disclosure and its moderators: a meta-analysis. Psychol Bull. 2006 Nov;132(6):823-65. doi: 10.1037/0033-2909.132.6.823. PMID 17073523
- [Background] Smyth JM, Stone AA, Hurewitz A, Kaell A. Effects of writing about stressful experiences on symptom reduction in patients with asthma or rheumatoid arthritis: a randomized trial. JAMA. 1999 Apr 14;281(14):1304-9. doi: 10.1001/jama.281.14.1304. PMID 10208146
- [Background] Pennebaker JW, Beall SK. Confronting a traumatic event: toward an understanding of inhibition and disease. J Abnorm Psychol. 1986 Aug;95(3):274-81. doi: 10.1037//0021-843x.95.3.274. No abstract available. PMID 3745650
- [Background] Andresen EM, Malmgren JA, Carter WB, Patrick DL. Screening for depression in well older adults: evaluation of a short form of the CES-D (Center for Epidemiologic Studies Depression Scale). Am J Prev Med. 1994 Mar-Apr;10(2):77-84. PMID 8037935
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- [Background] Weitzner MA, Jacobsen PB, Wagner H Jr, Friedland J, Cox C. The Caregiver Quality of Life Index-Cancer (CQOLC) scale: development and validation of an instrument to measure quality of life of the family caregiver of patients with cancer. Qual Life Res. 1999;8(1-2):55-63. doi: 10.1023/a:1026407010614. PMID 10457738
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Lee KC, Yiin JJ, Lu SH, Chao YF. The Burden of Caregiving and Sleep Disturbance Among Family Caregivers of Advanced Cancer Patients. Cancer Nurs. 2015 Jul-Aug;38(4):E10-8. doi: 10.1097/NCC.0000000000000166. PMID 24978619